CLINICAL TRIAL: NCT03643978
Title: A Randomized Controlled Trial of Decision Aids for Upper and Lower Extremity Conditions.
Brief Title: Decision Aids Upper and Lower Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care and Professor, Department of Surgery and Perioperative Care, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-07-0027
Record Dates: First submitted 2018-08-18; First posted 2018-08-23 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Upper Extremity Dysfunction; Lower Extremity Problem
Keywords: Decision aids
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in an intervention group that reviews a decision aid and a control group that does not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid Group (Experimental): These patients review a decision aid.
  Interventions: Other: Decision aid
- Control Group (No Intervention): These patients do not review a decision aid.

INTERVENTIONS:
Other: Decision aid — The decision aids aim to inform the patients about the diagnosis and the treatment options. They aim to help the patient prioritize and make an informed decision.
  Arms: Decision Aid Group

SUMMARY:
This study aims to assess differences in choice of treatment (and the rationale behind it), physical function, pain intensity, satisfaction, and decision regret between orthopedic patients who review a decision aid during their visit and those that do not. Decision aids for 23 different conditions are included.

DETAILED DESCRIPTION:
Patients visiting an orthopeadic surgeon in one of our 4 affiliated offices in a large urban area in the United States are invited to participate over a 4 month period. All English-speaking patients, between 18 and 89 years old, visiting an orthopeadic surgeon with a new problem, for which either invasive or non-invasive treatment is possible and a DA is available are asked to participate in this study. Exclusion criteria are non-English speakers or a clear preference for a treatment option by surgeon or patient. Patients will be randomly assigned to either the intervention or the control group in a 1:1 ratio using an Excel random number generator. Patients in the intervention group go over the DA during the visit, once the surgeon has identified the diagnosis. After the diagnosis is set, the surgeon steps out of the visit and steps back in when the patients has reviewed the DA. The surgeon and the patient go over the treatment options and a decision will be made. After the visit, all patients, both in the intervention and control group, are asked to fill out a survey. Two weeks after enrollment a research assistant calls all patients for a follow up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

English-speaking, adult patients seeing an upper or lower extremity surgeon for a new visit regarding diagnoses that can be treated invasively and non-invasively:

Shoulder

* Clavicle fracture in the middle
* Clavicle fracture close to the shoulder
* Proximal humerus fracture
* Humerus shaft fracture
* Distal humerus fracture

Elbow

* Lateral epicondylitis
* Ruptured biceps at the elbow
* Olecranon fracture
* Radial head fracture
* Olecranon bursitis

Hand/wrist

* Distal radius fracture
* Carpal tunnel syndrome
* Scaphoid fracture
* Thumb arthrosis
* Trigger finger
* Mallet fracture
* de Quervain tendinopathy
* Wrist ganglion
* Dupuytren

Knee • Knee arthritis: cortisone injection

Hip

• Hip arthritis: total hip arthroplasty

Exclusion Criteria:

* Obvious indication for one treatment approach, either from the surgeon or the patient perspective.
* Patients who do not want to be contacted for follow-up.
* Non-English speaking patients, because the decision aids used in this study are not currently validated to non-English language.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction on a 11-point ordinal scale | From enrollment till follow-up after two weeks
  On a scale of 0-10 how satisfied were you with this visit 0 being totally dissatisfied and 10 being totally satisfied.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Physical Function Computer Adaptive Test (directly after visit) | From enrollment till two weeks after visit
  Questionnaire that measures patients self-reported capability of physical activities.
  This Questionnaire is a CAT: Computerized Adaptive Test. Participant responses guide the system's choice of subsequent items from the full item bank (121 items in total in adult bank). Although items differ across respondents taking CAT, scores are comparable across participants.
  CAT will continue until either the standard error drops below a specified level, or the participant has answered the maximum number of questions (12), whichever occurs first.
  A score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. Range scores 19-76. Higher scores is better physical function.
Pain intensity on an 11-point ordinal scale | From enrollment till two weeks after visit
  Can you rate your pain on a scale of 0-10, 0 meaning no pain and 10 meaning the worst possible pain.
Decision regret scale (O'Connor '96) | One time measurement, two weeks after the visit.
  Measures 'distress' or 'remorse' after a (health care) decision. Scale from 1-5, 1 being strongly agree, 5 being stongly disagree
  1. it was the right decision
  2. I regret the choice that was made
  3. I would go for the same chice if I had to do it over again
  4. The choice did me a lot of harm
  5. The decision was a wise one
Choice of treatment (invasive/non-invasive) | Day of enrollment
  Patients have to fill out if they either chose invasive treatment (surgery) or non-invasive treatment (no surgery)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Austin Regional Clinic, Austin, Texas
  - Texas Orthopedics, Austin, Texas
  - HTB Musculoskeletal Institute, Austin, Texas
  - Seton Institute for Plastic and Reconstructive Surgery, Austin, Texas
  - Orthopedic Specialists of Austin, Austin, Texas
  - ATX Ortho, Austin, Texas

IPD SHARING:
Plan to Share IPD: No